CLINICAL TRIAL: NCT03203421
Title: A Phase I/II Study to Assess the Safety, Immunogenicity and Protective Efficacy of Novel Malaria Vaccine Candidates ChAdOx1 LS2 and MVA LS2 in Healthy UK Adults
Brief Title: A Safety and Efficacy Study of ChAdOx1 LS2 and MVA LS2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VAC067
Record Dates: First submitted 2017-06-27; First posted 2017-06-29 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2017-08

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low Dose (Group 1) (Active Comparator): One low dose of ChAdOx1 LS2 (5 x 10^9 vp) on day 0.
  Interventions: Biological: ChAdOx1 LS2
- Prime-Boost (Group 2) (Active Comparator): One high dose of ChAdOx1 LS2 (2.5 x 10^10 vp) on day 0 and one dose of MVA LS2 (2 x 10^8 pfu) on day 56.
  Interventions: Biological: ChAdOx1 LS2; Biological: MVA LS2
- Control Group A (No Intervention): No vaccinations will be administered.
- Control Group B (No Intervention): No vaccinations will be administered.

INTERVENTIONS:
Biological: ChAdOx1 LS2 — A viral vectored vaccine, using a chimpanzee adenovirus as a vector encoding malaria liver-stage dual antigen LS2 (LSA1 and LSAP2) fused with the transmembrane domain from shark invariant chain.
  Arms: Low Dose (Group 1); Prime-Boost (Group 2)
Biological: MVA LS2 — Modified vaccinia Ankara vector encoding liver-stage dual antigen LS2 (LSA1 ad LSAP2) fused to the C-terminal end of the leader sequence of tPA.
  Arms: Prime-Boost (Group 2)

SUMMARY:
The purpose of this study is to assess the safety, immunogenicity and efficacy of the candidate malaria vaccines ChAdOx1 LS2 and MVA LS2.

Healthy adult volunteers will be recruited and vaccinated in Oxford.

DETAILED DESCRIPTION:
This is an open label, dose-escalation, first in human, partially blinded, phase I/IIa controlled human malaria infection (CHMI) study. The study will assess the safety, immunogenicity and protective efficacy of the novel malaria vaccine candidates ChAdOx1 LS2 and MVA LS2 in healthy UK adults.

Healthy, malaria naive adults, aged between 18 and 45 years, will be recruited and vaccinated in Oxford.

A total of between 23 and 31 volunteers will be recruited across four groups:

Group 1 volunteers will receive a low dose ChAdOx1 LS2 vaccination on day 0. Group 2 volunteers will receive a high dose ChAdOx1 LS2 vaccination on day 0 and a dose of MVA LS2 on day 56, followed by a CHMI on day 77. Volunteers exhibiting sterile protection will undergo a repeat CHMI 5-7 months later.

Control Group A will not receive any vaccinations and will undergo CHMI on day 77.

Control Group B will not receive any vaccinations and will undergo CHMI during the repeat challenge.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 45 years
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner
* For females only, willingness to practice continuous effective contraception (see below) during the study and a negative pregnancy test on the day(s) of screening and vaccination
* Agreement to refrain from blood donation during the course of the study
* Provide written informed consent to participate in the trial.

Additional inclusion criteria for group 2 and control groups A&B:

* Agreement to refrain from blood donation during the course of the study and for at least 3 years after the end of their involvement in the study.
* Reachable (24/7) by mobile phone during the period between CHMI and completion of antimalarial treatment.
* Willingness to take a curative anti-malaria regimen following CHMI.
* For volunteers not living in Oxford: agreement to stay in a hotel room close to the trial centre during a part of the study (from at least day 6.5 post mosquito bite until anti-malarial treatment is completed).
* Answer all questions on the informed consent quiz correctly.

Exclusion Criteria:

* History of clinical malaria (any species).
* Travel to a clearly malaria endemic locality during the study period or within the preceding six months
* Receipt of an investigational product in the 30 days preceding enrolment, or planned receipt during the study period.
* Prior receipt of an investigational vaccine likely to impact on interpretation of the trial data as assessed by the investigator. This may include non-malaria adenovirus vectored experimental vaccine. If any volunteers in Group 2 undergo rechallenge, this exclusion criterion does not extend to the vaccines previously received in the VAC067 trial.
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed).
* Use of immunoglobulins or blood products within 3 months prior to enrolment.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine (e.g. egg products, Kathon) or malaria infection.
* Any history of anaphylaxis post vaccination.
* History of clinically significant contact dermatitis.
* Pregnancy, lactation or intention to become pregnant during the study.
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* History of serious psychiatric condition that may affect participation in the study.
* Any other serious chronic illness requiring hospital specialist supervision.
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 standard UK units every week.
* Suspected or known injecting drug abuse in the 5 years preceding enrolment.
* Hepatitis B surface antigen (HBsAg) detected in serum.
* Seropositive for hepatitis C virus (antibodies to HCV) at screening (unless has taken part in a prior hepatitis C vaccine study with confirmed negative HCV antibodies prior to participation in that study, and negative HCV RNA PCR at screening for this study).
* Inability of the study team to contact the volunteer's GP to confirm medical history and safety to participate
* Any clinically significant abnormal finding on biochemistry or haematology blood tests, urinalysis or clinical examination. In the event of abnormal test results, confirmatory repeat tests will be requested (described in section 9.6.1).
* Any other significant disease, disorder, or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.

Additional exclusion criteria for group 2 and control groups A&B:

* Clinically significant disturbances of electrolyte balance, eg, hypokalaemia or hypomagnesaemia
* Use of systemic antibiotics with known antimalarial activity within 30 days of CHMI (e.g. trimethoprim-sulfamethoxazole, doxycycline, tetracycline, clindamycin, erythromycin, fluoroquinolones and azithromycin).
* History of sickle cell anaemia, sickle cell trait, thalassaemia or thalassaemia trait or any haematological condition that could affect susceptibility to malaria infection.
* Use of medications known to cause prolongation of the QT interval and existing contraindication to the use of Malarone.
* Use of medications known to have a potentially clinically significant interaction with Riamet and Malarone.
* Contraindications to the use of both Riamet and Malarone.
* Any clinical condition known to prolong the QT interval and existing contraindication to the use of Malarone.
* Family history of congenital QT prolongation or sudden death and existing contraindication to the use of Malarone.
* History of cardiac arrhythmia, including clinically relevant bradycardia and existing contraindication to the use of Malarone.
* Positive family history in both 1st and 2nd degree relatives < 50 years old for cardiac disease.
* Volunteer unable to be closely followed for social, geographic or psychological reason.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of ChAdOx1 LS2 administered alone and with MVA LS2 in a prime-boost vaccination regimen in healthy malaria-naive volunteers assessed by the frequency and severity of adverse events. | 31 - 40 weeks
  The number of participants who experience adverse events and the severity of any adverse events.
The efficacy of ChAdOx2 LS2 and MVA LS2 administered in a prime-boost vaccination regimen against malaria sporozoite challenge, in healthy malaria-naive volunteers. | 90 days
  The occurrence of Plasmodium falciparum parasitemia, assessed by blood slide and polymerase chain reaction (PCR).

CONTACTS AND LOCATIONS:
Locations (1):
- CCVTM, University of Oxford, Churchill Hospital, Oxford, United Kingdom